CLINICAL TRIAL: NCT00624702
Title: A Multi-center, Randomized, Single-dose, Double-blind, 4-way Cross-over Study to Evaluate Tolerability Following Treatment With Indacaterol Salts (Maleate, Xinafoate and Acetate) in Comparison to Placebo in Patients With Mild to Moderate Persistent Asthma
Brief Title: Tolerability of Indacaterol Salts (Maleate, Xinafoate and Acetate) in Comparison to Placebo in Patients With Mild to Moderate Persistent Asthma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Novartis, Novartis
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CQAB149B2102
Record Dates: First submitted 2008-02-15; First posted 2008-02-27 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2010-08

CONDITIONS: Asthma
Keywords: Asthma, cough, spirometry, maleate, xinafoate, acetate, SDDPI (single dose dry powder inhaler)
MeSH Terms: conditions — Asthma; Cough

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): Active Comparator 1 different salt formulation of Indacaterol.
  Interventions: Drug: Indacaterol maleate
- 2 (Active Comparator): Active Comparator 2 different salt formulation of Indacaterol.
  Interventions: Drug: Indacaterol maleate
- 3 (Active Comparator): Active Comparator 3 different salt formulation of Indacaterol.
  Interventions: Drug: Indacaterol maleate
- 4 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Indacaterol maleate — Four single dose treatments (each dose is 400 µg-for the active salts-via SDDPI), with at least a 7 day inter-dose interval
  Arms: 1
Drug: Indacaterol maleate — Four single dose treatments (each dose is 400 µg-for the active salts-via SDDPI), with at least a 7 day inter-dose interval
  Arms: 2
Drug: Indacaterol maleate — Four single dose treatments (each dose is 400 µg-for the active salts-via SDDPI), with at least a 7 day inter-dose interval
  Arms: 3
Drug: Placebo
  Arms: 4

SUMMARY:
This study will explore information on whether changing the salt formulation of indacaterol affects the incidence of post-inhalation cough.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients 18 to 65 years old (inclusive)
* Patients with mild to moderate persistent asthma
* BMI must be within the range of 18-32 kg/m2 inclusive
* Female subjects must:

  1. have been sterilized at least 6 months prior to screening
  2. be post-menopausal with no regular bleeding for at least a year prior to inclusion

Exclusion Criteria:

* Patients with life-threatening arrhythmias
* Patients with COPD or diabetes mellitus
* History of immunocompromise, including a positive HIV
* A positive Hepatitis B surface antigen (HBsAg) of Hepatitis C test result

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2008-02; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Presence of cough within 5 minutes post dose and the onset of cough (relative to inhalation) | throughout the study
Severity of cough: to be judged independently by both the patient and the physician | throughout the study
Occurrence of cough within 1 minute post dose | throughout the study
Number of coughs | throughout the study
Duration of coughing | throughout the study

SECONDARY OUTCOMES:
Presence of cough within 5 minutes post dose and the onset of cough (relative to inhalation) | throughout the study
Severity of cough: to be judged independently by both the patient and the physician | throughout the study
Occurrence of cough within 1 minute post dose | throughout the study
Number of coughs | throughout the study
Duration of coughing | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Novartis investigator site
Locations (2):
- Canada (2):
  - Novartis Investigator Site, Ottawa, Ontario
  - Novartis Investigator Site, Montreal, Quebec

REFERENCES:
- See also: Results for QAB149B2102 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=3022